CLINICAL TRIAL: NCT05685173
Title: A Phase 1 Study to Assess Safety and Tolerability of REGN5837, an Anti-CD22 x Anti-CD28 Costimulatory Bispecific Monoclonal Antibody, in Combination With Odronextamab, an Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody, in Patients With Aggressive B-Cell Non-Hodgkin Lymphomas (ATHENA-1)
Brief Title: A Trial to Study if REGN5837 in Combination With Odronextamab is Safe for Adult Participants With Aggressive B-cell Non-Hodgkin Lymphomas
Acronym: ATHENA-1
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R5837-ONC-2019; 2020-005084-32 (EudraCT Number); 2022-502137-26-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2022-12-14; First posted 2023-01-13 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: B-cell Non-Hodgkins Lymphoma (B-NHL)
Keywords: Aggressive B-Cell Non-Hodgkin Lymphomas; Relapsed or Refractory
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Odronextamab and REGN5837 (Experimental): Odronextamab and REGN5837 will be administered by IV infusion using a step-up dosing schedule.
  Interventions: Drug: Odronextamab; Drug: REGN5837

INTERVENTIONS:
Drug: Odronextamab — Odronextamab will be administered by IV infusion
  Other Names: REGN1979
Drug: REGN5837 — REGN5837 will be administered by IV infusion

SUMMARY:
The study is researching an experimental drug called REGN5837 in combination with another experimental drug, odronextamab (called "study drugs").

The aim of the study is to see how safe and tolerable the study drugs are, and to define the recommended dose for phase 2.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How much study drug is in the blood at different times
* Whether the body makes antibodies against the study drugs (that could make the drugs less effective or could lead to side effects)
* To find out how well the study drugs work against relapsed or refractory aggressive B-cell non-Hodgkin lymphomas (B-NHLs)

ELIGIBILITY:
Key Inclusion Criteria:

1. Have documented CD20+ aggressive B-NHL, with disease that has progressed after at least 2 lines of systemic therapy containing an anti-CD20 antibody and an alkylating agent, as described in the protocol.
2. Measurable disease on cross sectional imaging as defined in the protocol
3. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
4. Adequate bone marrow, renal and hepatic function as defined in the protocol
5. Availability of tumor tissue for submission to central laboratory is required for study enrollment. Archival tumor tissue for histological assessment prior to enrollment is allowed
6. During dose expansion phase of the study, participant should be willing to undergo mandatory tumor biopsies, if in the opinion of the investigator, the participant has an accessible lesion that can be biopsied without significant risk to the participant.

Key Exclusion Criteria:

1. Prior treatments with allogeneic stem cell transplantation or solid organ transplantation, treatment with anti-CD20 x anti- CD3 bispecific antibody, such as odronextamab
2. Diagnosis of mantle cell lymphoma (MCL)
3. Primary central nervous system (CNS) lymphoma or known involvement by non-primary CNS lymphoma, as described in the protocol
4. Treatment with any systemic anti-lymphoma therapy within 5 half-lives or within 14 days prior to first administration of study drug, whichever is shorter, as described in the protocol
5. Standard radiotherapy within 14 days of first administration of study drug, as described in the protocol
6. Continuous systemic corticosteroid treatment with more than 10 mg per day of prednisone or corticosteroid equivalent within 72 hours of start of odronextamab
7. Co-morbid conditions, as described in the protocol
8. Infections, as described in the protocol
9. Allergy/hypersensitivity: Known hypersensitivity to both allopurinol and rasburicase

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2027-06-02 (Estimated); Study Completion 2029-05-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) of REGN5837 in combination with odronextamab | From Cycle 2, Day 15 to Cycle 4, Day 7 (each induction cycle is 21 days)
  A DLT is defined as any non-haematologic and haematologic toxicity, as defined in the protocol, unless the event is clearly attributable to the underlying disease or to an extraneous cause (including concomitant medications).
Incidence of treatment-emergent adverse events (TEAEs) of REGN5837 in combination with odronextamab | Up to approximatively 5 years
  Treatment-emergent adverse events (TEAEs) are defined as those AEs that newly occurred or worsened during the on-treatment period and any treatment-related serious adverse events (SAEs) that occurred during the post-treatment period.
Severity of TEAEs of REGN5837 in combination with odronextamab | Up to approximatively 5 years
  Treatment-emergent adverse events (TEAEs) are defined as those AEs that newly occurred or worsened during the on-treatment period and any treatment-related serious adverse events (SAEs) that occurred during the post-treatment period.
Incidence of adverse events of special interest (AESIs) of REGN5837 in combination with odronextamab | Up to approximatively 5 years
  An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate.
Severity of AESIs of REGN5837 in combination with odronextamab | Up to approximatively 5 years
  An AESI (serious or non-serious) is one of scientific and medical concern specific to the sponsor's product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate.

SECONDARY OUTCOMES:
Concentrations of REGN5837 in the serum | Up to 90 days post last study drug administration
Concentrations of odronextamab in the serum | Up to 90 days post last study drug administration
Incidence of anti-drug antibodies (ADAs) to REGN5837 over the study duration | Up to 90 days post last study drug administration
Incidence of ADAs to odronextamab over the study duration | Up to 90 days post last study drug administration
Titer of ADAs to REGN5837 over the study duration | Up to 90 days post last study drug administration
Titer of ADAs to odronextamab over the study duration | Up to 90 days post last study drug administration
Overall response rate (ORR) according to the Lugano Classification of response | Up to approximatively 5 years
  The ORR is defined as the proportion of patients who achieve a best overall response CR or PR during or following study treatment according to the Lugano Classification based on local investigator review.
Complete response (CR) rate according to the Lugano Classification of response | Up to approximatively 5 years
  The CR rate is defined as the proportion of patients who achieve a best overall response CR during or following study treatment according to the Lugano Classification based on local investigator review.
Progression free survival (PFS) according to the Lugano Classification of response | Up to approximatively 5 years
  PFS is defined as the time from the start of study treatment until the first date of progressive disease, or death due to any cause, whichever occurs first, based on local investigator review.
Overall survival (OS) | Up to approximatively 5 years
  OS is measured from the start of study treatment until death due to any cause.
Duration of Response (DoR) according to the Lugano Classification of response | Up to approximatively 5 years
  DOR is defined for responders (patients with a best overall response of CR or PR). It is the time from the date of the first documented CR or PR until the date of the first date of progressive disease, or death due to any cause, whichever occurs first, based on local investigator review.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (20):
- United States (9):
  - City of Hope, Duarte, California
  - University of California Los Angeles (UCLA) Medical Center, Santa Monica, California
  - Norton Cancer Institute, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard Medical School - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Health Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - UT Southwestern, Dallas, Texas
- France (3):
  - CHU de Bordeaux, Talence, Nouvelle-Aquitaine
  - Hopital Saint Louis, Paris, Paris
  - Gustave Roussy, Villejuif, Île-de-France Region
- Netherlands (2):
  - Erasmus Medical Center Rotterdam, Rotterdam, South Holland
  - Amsterdam University Medical Centre, location AMC, Amsterdam
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - University Hospital and Research Institute, Madrid, Madrid
- United Kingdom (4):
  - Royal Cornwall Hospital NHS Trust, Truro, Cornwall
  - Southampton General Hospital, Southampton, Hampshire
  - The Christie NHS Foundation Trust, Manchester, Manchester
  - Western General Hospital, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli.
  Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/